CLINICAL TRIAL: NCT01524029
Title: Digital Breast Tomosynthesis vs. Digital Mammography: A National Multicenter Trial
Brief Title: Digital Breast Tomosynthesis Versus Digital Mammography: A National Multicenter Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Moritz, Assistenzarzt, Medical University of Vienna
Other Study IDs: TomoTrial001
Record Dates: First submitted 2012-01-29; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Breast Neoplasms
Keywords: Digital Breast Tomosynthesis; Digital Mammography; Breast cancer detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast Cancer Screening Patients: Group 1 consists of Women referred to Breast Cancer Screening examinations at a participating Austrian Breast Imaging Site
- Diagnostic Patients: Patients referred to a participating Breast Imaging Center for a clinically or radiologically detected breast lesion

SUMMARY:
The goal of this study is to determine the value of the new mammography technique called Digital Breast Tomosynthesis (DBT) compared to the current standard technique Digital Mammography for the early detection of Breast Cancer.

DBT is able to compute a three-dimensional image of a breast from several low-dose mammographies taken from different angles while the device is moving around the breast in a circular motion. This should overcome a significant limitation of Digital Mammography arising from the masking of breast cancer in a mammography image caused by overlying normal breast tissue.

This is a study conducted in several Austrian Breast Imaging Centers.

DETAILED DESCRIPTION:
This prospective national multicenter multivendor trial aims at determining the impact of the novel technique Digital Breast Tomosynthesis (DBT) in the assessment and screening for breast cancer. Mammography is the primary imaging modality for the early detection of clinically occult breast cancer.

Despite advances in mammographic technique, mammography is still limited with regard to both sensitivity and specificity. In the majority of cases these limitations arise from the masking of subtle breast cancer lesions by overlapping breast tissue.

DBT is a novel technique that tries to overcome these limitations by performing a 3D-reconstruction of breast tissue from multiple low-dose digital mammographic images acquired in several planes in a 15 to 50 degree angle.

Early studies indicate an advantage of DBT compared to the standard Full Field Digital Mammography (FFDM) in terms of an improvement of specificity without cutback in sensitivity.

Controversy continues over the use of DBT in combination with FFDM or as a standalone screening method without concomitant 2D imaging. Unfortunately, the peer-reviewed publications evaluating DBT are limited and consist of single institution studies with a small number of participants.

The purpose of this study is to evaluate the novel technique of DBT compared to routine FFDM in a clinical large sample study (600 participants) to provide the path to implementation of this new technique into clinical and screening routine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 25 years (40 years or older for Screening Cohort)
* No history of breast cancer
* Written informed consent
* Asymptomatic women in follow up for early detection of breast cancer or
* Patients with a recent positive mammography (BI-RADS 3-5)

Exclusion Criteria:

* Pregnant and breast feeding women
* Unable to tolerate breast compression
* Breast implants
* Unable to understand or execute written informed consent

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of two groups:
  One screening group consisting of asymptomatic women (Age 40+) referred for a screening mammography examination.
  The second group consists of women aged 25+ referred for further examination of a breast lesion.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Specificity of Digital Breast Tomosynthesis in the characterization of Breast lesions | One year

SECONDARY OUTCOMES:
Sensitivity of Digital Breast Tomosynthesis in the detection of malignant breast lesions | One year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Moritz, MD, Principal Investigator — Medical University of Vienna; Thomas Helbich, MD Prof. MBA MSc, Study Director — Medical University of Vienna
Locations (5):
- Austria (5):
  - Medical University of Graz, Graz, Styria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - Medical University of Vienna, Vienna
  - Kaiser Franz Josef Spital, Vienna
  - Hanusch Krankenhaus, Vienna